CLINICAL TRIAL: NCT01257737
Title: Long Term Use of HPN-100 in Urea Cycle Disorders
Brief Title: To Evaluate the Safety of Long-term Use of HPN-100 in the Management of Urea Cycle Disorders (UCDs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPN-100-011
Record Dates: First submitted 2010-12-02; First posted 2010-12-10 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Disorders; GT4P; HPN-100; Sodium Phenylbutyrate (NaPBA); Glyceryl tri-(4-phenylbutyrate); Phenylbutyrate; Hyperion; BUPHENYL; hyperammonemia
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HPN-100 (Experimental): Participants continued HPN-100 treatment after completion of HPN-100-005SE, HPN-100-007, or HPN-100-012SE.
  Interventions: Drug: HPN-100

INTERVENTIONS:
Drug: HPN-100 — Participants received individualized doses of HPN-100 orally, three times daily (TID) with meals. The initial dose was the same dose administered at the end of the HPN-100-005SE, HPN-100-007, or HPN-100-012SE studies. Dose adjustments (including frequency adjustments) were permitted as judged clinically appropriate by the investigator based on assessment of ammonia-scavenging needs (e.g., severity of the UCD defect, dietary protein intake, and urinary phenylacetylglutamine [PAGN] excretion). The maximum recommended dose of HPN-100 in participants weighing less than 20 kg was 0.53 mL/kg/day (equivalent to 600 mg/kg/day of NaPBA), and was 11.48 mL/m²/day in heavier subjects (equivalent to 13g/m²/day of NaPBA). The maximum HPN-100 dose recommended per protocol was 17.4 mL/day, which is equivalent to 20 g/day of NaPBA.
  Other Names: GT4P, Glyceryl tri-(4-phenylbutyrate), RAVICTI

SUMMARY:
This was an open-label, long-term safety study of HPN-100 (RAVICTI; glycerol phenylbutyrate) in participants with a urea cycle disorder (UCD) who completed the safety extensions of HPN-100-005 (NCT00947544; HPN-100-005SE), HPN-100-006 (NCT00947297; HPN-100-007), or HPN-100-012 (NCT01347073; HPN-100-012SE). The initial studies were 1- to 2-week crossover studies, and their associated safety extensions were 12-month, open-label studies. All participants who completed the initial studies were eligible to enroll in the associated safety extension studies, and new participants were also permitted to enroll directly into the safety extension studies.

DETAILED DESCRIPTION:
The duration of treatment in this study was open-ended. Participants were to return for clinic visits as prescribed by the investigator, and were to be seen at a minimum of every 6 months. At each clinic visit, participants were queried about any adverse events (AEs) or hyperammonemic crises (HACs) that occurred since the last visit. Physical and neurological examinations were performed, and blood samples were collected for the analysis of ammonia, amino acid panels, and routine clinical laboratory safety tests. Participants underwent neuropsychological testing at baseline, every 12 months thereafter, and at the final study visit.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who completed Studies HPN-100-005SE, HPN-100-007, or HPN-100-012SE
* Signed informed consent by participant and/or participant's legally authorized representative
* Negative pregnancy test for all females of childbearing potential

Exclusion Criteria:

* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may have put the participant at increased risk when participating
* Known hypersensitivity to PAA (phenylacetate) or PBA (phenylbutyrate).
* Liver transplant, including hepatocellular transplant
* Pregnant, breastfeeding or lactating females

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-10-04 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- United States (15):
  - UCLA Pediatrics/Genetics, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Denver Children's Hospital, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Maine Medical Center, Portland, Maine
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Pittsburg of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Groups:
- HPN-100- Pediatric: Pediatric participants (age 1-17) continued HPN-100 treatment after completion of HPN-100-005SE, HPN-100-007, or HPN-100-012SE.
- HPN-100 - Adult: Adult participants (age 19-61) continued HPN-100 treatment after completion of HPN-100-005SE, HPN-100-007, or HPN-100-012SE.
Period: Overall Study
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
Started | 45 | 43
Completed | 43 | 39
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Liver transplant | 1 | 0
Not completed — Relocation out of the country | 0 | 1
Not completed — Withdrew from study | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received any amount of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (4.33) | 33.3 (11.90) | 20.0 (15.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 13 | 17 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 38 | 36 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Urea Cycle Disorder Diagnosis [Count of Participants; unit: Participants]
  Argininosuccinate synthetase (ASS) deficiency | 7 | 2 | 9
  Ornithine transcarbamylase (OTC) deficiency | 26 | 35 | 61
  Arginase (ARG) deficiency | 1 | 1 | 2
  Argininosuccinate lyase (ASL) deficiency | 11 | 2 | 13
  Hyperornithinemia-hyperammonemia-homocitrullinuria | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: Safety was assessed by the incidence of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs). An AE/adverse experience was any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. For additional information regarding adverse events, please see the safety section of the record.
Time Frame: From the time of informed consent until 7 days after the last dose of study drug, up to 66 months
Population: Safety Population: All participants who received any amount of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
Number analyzed (Participants) | 45 | 43
Participants | 34 | 40

2. Secondary Outcome: Mean Normalized Blood Ammonia Levels
Description: Blood samples were collected for the assessment of plasma ammonia concentrations at baseline, at least every 6 months, at all unscheduled visits, and at the end of study participation. Ammonia level data were obtained from different local laboratories and each laboratory may have used a slightly different normal reference range. Therefore, the ammonia level data were normalized to a standard laboratory reference range before performing any analysis of ammonia data.
Time Frame: From baseline through the end of the study, up to 66 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
Number analyzed (Participants) | 44 | 43
μmol/L
  Baseline | 19.445 (16.4478) | 26.005 (23.4156)
  Month 6: number analyzed (Participants) | 25 | 38
  Month 6 | 18.437 (14.7127) | 24.235 (18.2070)
  Month 12: number analyzed (Participants) | 23 | 38
  Month 12 | 18.236 (13.7955) | 27.843 (20.3701)
  Month 18: number analyzed (Participants) | 23 | 39
  Month 18 | 25.145 (26.2123) | 31.378 (26.1624)
  Month 24: number analyzed (Participants) | 11 | 13
  Month 24 | 15.428 (11.8506) | 26.044 (12.5713)
  Month 30: number analyzed (Participants) | 2 | 4
  Month 30 | 19.139 (15.1512) | 31.140 (21.6156)
  Month 36: number analyzed (Participants) | 1 | 4
  Month 36 | 9.265 | 39.890 (31.2392)
  Month 42: number analyzed (Participants) | 1 | 4
  Month 42 | 10.294 | 21.360 (9.1448)
  Month 48: number analyzed (Participants) | 1 | 4
  Month 48 | 53.529 | 15.956 (7.9071)
  Month 54: number analyzed (Participants) | 1 | 4
  Month 54 | 42.206 | 45.810 (25.5722)
  Month 60: number analyzed (Participants) | 1 | 4
  Month 60 | 42.21 | 50.175 (52.9026)
  Month 66: number analyzed (Participants) | 1 | 1
  Month 66 | 9.26 | 9.26
  End of Study: number analyzed (Participants) | 39 | 33
  End of Study | 20.412 (14.4513) | 32.340 (31.2273)

3. Secondary Outcome: Number of Hyperammonemic Crises
Description: An hyperammonemic crisis (HAC) was defined as clinical symptoms associated with a venous ammonia concentration of ≥100 μmol/L.
Time Frame: From the time of informed consent until 7 days after the last dose of study drug, up to 66 months
Population: Safety Population: All participants who received any amount of study medication
Measure: Number; unit: Number of crises
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
Number analyzed (Participants) | 45 | 43
Number of crises | 22 | 22

4. Secondary Outcome: Causes of Hyperammonemic Crises
Description: An hyperammonemic crisis (HAC) was defined as clinical symptoms associated with a venous ammonia concentration of ≥100 μmol/L. Peak observed ammonia concentrations during an HAC, precipitating factors, and symptoms recorded as suggestive to hyperammonemia were documented. There can be multiple contributing factors to an hyperammonemic crisis; in some cases several causes were identified.
Time Frame: From the time of informed consent until 7 days after the last dose of study drug, up to 66 months
Population: Participants who experienced hyperammonemic crises
Measure: Number; unit: Number of crises
Units Other Than Participants: Hyperammonemic crises
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
Number analyzed (Participants) | 11 | 10
Number analyzed (Hyperammonemic crises) | 22 | 22
Number of crises
  Change in Diet | 0 | 4
  Non-compliance with urea cycle disorder medication | 1 | 0
  Infection | 6 | 0
  Intercurrent illness | 6 | 4
  Non-compliance with study drug | 2 | 4
  Unknown | 4 | 4
  Other | 5 | 9
  None | 1 | 4

5. Secondary Outcome: Mean Wechsler Abbreviated Scale of Intelligence (WASI) Scores
Description: The Wechsler Abbreviated Scale of Intelligence (WASI) was administered to adults and pediatric participants who were at least 6 years of age. It was used to estimate general intellectual ability (IQ) based on the vocabulary and matrix reasoning subtests. The vocabulary subtest included 4 images and 38 verbal items. In the matrix reasoning subtest, the participant viewed 35 incomplete grid patterns and was asked to complete the pattern using responses from 5 possible choices. The number of correct responses for each of the subtests was converted to a T-score using the WASI assessment manual; T-scores are standard scores with a mean of 50 and a standard deviation (SD) of 10. Raw scores for the 2 subtests were summed, and converted to a standard score (mean of 100 with SD of 15) for the general IQ score for adults and to a T-score for children in accordance with the WASI manual. Higher scores indicate a higher level of intelligence.
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and study exit visit (up to 66 months)
Population: Participants ≥ 6 years of age with available data; data were not analyzed for the 5 ongoing participants in Canada after the cutoff for the clinical study report (29 Oct 2015).
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
Number analyzed (Participants) | 28 | 41
T-score
  Vocabulary T Score- Baseline | 46.5 (13.53) | 45.2 (14.43)
  Vocabulary T Score- Month 12: number analyzed (Participants) | 24 | 35
  Vocabulary T Score- Month 12 | 48.9 (11.66) | 44.2 (15.59)
  Vocabulary T Score- Month 24: number analyzed (Participants) | 9 | 12
  Vocabulary T Score- Month 24 | 44.9 (12.48) | 45.2 (13.99)
  Vocabulary T Score- Month 36: number analyzed (Participants) | 1 | 2
  Vocabulary T Score- Month 36 | 20.0 | 36.5 (23.33)
  Vocabulary T Score- Month 48: number analyzed (Participants) | 1 | 1
  Vocabulary T Score- Month 48 | 20.0 | 20.0
  Vocabulary T Score- Study Exit: number analyzed (Participants) | 24 | 36
  Vocabulary T Score- Study Exit | 47.8 (11.42) | 44.3 (15.87)
  Matrix Reasoning T Score- Baseline: number analyzed (Participants) | 27 | 41
  Matrix Reasoning T Score- Baseline | 46.8 (10.37) | 45.5 (15.24)
  Matrix Reasoning T Score- Month 12: number analyzed (Participants) | 24 | 35
  Matrix Reasoning T Score- Month 12 | 48.8 (12.91) | 46.5 (15.88)
  Matrix Reasoning T Score- Month 24: number analyzed (Participants) | 9 | 12
  Matrix Reasoning T Score- Month 24 | 50.0 (14.82) | 48.0 (16.75)
  Matrix Reasoning T Score- Month 36: number analyzed (Participants) | 1 | 2
  Matrix Reasoning T Score- Month 36 | 20.0 | 44.5 (24.75)
  Matrix Reasoning T Score- Month 48: number analyzed (Participants) | 1 | 1
  Matrix Reasoning T Score- Month 48 | 20.0 | 25.0
  Matrix Reasoning T Score- Study Exit: number analyzed (Participants) | 24 | 36
  Matrix Reasoning T Score- Study Exit | 49.2 (12.53) | 46.1 (16.07)
  Est. Full Scale IQ T Score- Baseline: number analyzed (Participants) | 27 | 0
  Est. Full Scale IQ T Score- Baseline | 95.6 (17.07) |
  Est. Full Scale IQ T Score- Month 12: number analyzed (Participants) | 22 | 0
  Est. Full Scale IQ T Score- Month 12 | 99.5 (18.72) |
  Est. Full Scale IQ T Score- Month 24: number analyzed (Participants) | 8 | 0
  Est. Full Scale IQ T Score- Month 24 | 97.5 (21.58) |
  Est. Full Scale IQ T Score- Month 36: number analyzed (Participants) | 1 | 0
  Est. Full Scale IQ T Score- Month 36 | 55 |
  Est. Full Scale IQ T Score- Study Exit: number analyzed (Participants) | 22 | 0
  Est. Full Scale IQ T Score- Study Exit | 99.5 (18.18) |
  Est. Full Scale IQ Standard Score- Baseline: number analyzed (Participants) | 0 | 41
  Est. Full Scale IQ Standard Score- Baseline |  | 95.1 (20.85)
  Est. Full Scale IQ Standard Score- Month 12: number analyzed (Participants) | 2 | 35
  Est. Full Scale IQ Standard Score- Month 12 | 92.0 (8.49) | 93.9 (22.61)
  Est. Full Scale IQ Standard Score- Month 24: number analyzed (Participants) | 1 | 12
  Est. Full Scale IQ Standard Score- Month 24 | 97.0 | 94.7 (24.03)
  Est. Full Scale IQ Standard Score- Month 36: number analyzed (Participants) | 0 | 2
  Est. Full Scale IQ Standard Score- Month 36 |  | 85.5 (33.23)
  Est. Full Scale IQ Standard Score- Month 48: number analyzed (Participants) | 1 | 1
  Est. Full Scale IQ Standard Score- Month 48 | 51.0 | 55.0
  Est. Full Scale IQ Standard Score- Study Exit: number analyzed (Participants) | 4 | 36
  Est. Full Scale IQ Standard Score- Study Exit | 85.5 (24.69) | 93.5 (23.24)

6. Secondary Outcome: Mean Child Behavior Checklist (CBCL) Problems Scores
Description: The Child Behavior Checklist (CBCL) is a widely-used method of identifying problem behavior. Two versions of the CBCL were used in this study; the assessment for children 6-18 years of age was used for participants ≥6 years of age, and the assessment for children 1.5-5 years of age was used for those who were at least 5 years old but <6 years of age. Parents/caregivers answered questions (120 and 100 questions, respectively, for the older and younger populations) using a 3-point Likert scale (0= not true; 1= somewhat or sometimes true; 2 =very true or often true). Using a computer program, responses to similar questions were grouped together into 20 domains (e.g., activities, social, school, etc.), and domain response scores were converted to T-scores and percentiles. A mean score of 50 is average, with a standard deviation of 10 points. Higher scores indicate greater problems. The total problems score is the sum of all of the problem items.
Time Frame: Baseline, Month 12, Month 24, and study exit visit (up to 66 months)
Population: Participants 5-18 years of age with available data; data were not analyzed for the 1 ongoing pediatric participant in Canada after the cutoff for the clinical study report (29 Oct 2015).
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | HPN-100- Pediatric
Number analyzed (Participants) | 31
T-Score
  Internalizing Problems T Score- Baseline | 53.4 (14.01)
  Internalizing Problems T Score- Month 12: number analyzed (Participants) | 21
  Internalizing Problems T Score- Month 12 | 52.5 (13.88)
  Internalizing Problems T Score- Month 24: number analyzed (Participants) | 6
  Internalizing Problems T Score- Month 24 | 55.5 (11.61)
  Internalizing Problems T Score- Study Exit: number analyzed (Participants) | 21
  Internalizing Problems T Score- Study Exit | 52.5 (13.22)
  Externalizing Problems T Score- Baseline | 53.5 (13.19)
  Externalizing Problems T Score- Month 12: number analyzed (Participants) | 21
  Externalizing Problems T Score- Month 12 | 52.1 (10.51)
  Externalizing Problems T Score- Month 24: number analyzed (Participants) | 6
  Externalizing Problems T Score- Month 24 | 54.8 (9.68)
  Externalizing Problems T Score- Study Exit: number analyzed (Participants) | 21
  Externalizing Problems T Score- Study Exit | 53.0 (10.30)
  Affective Problems T Score- Baseline: number analyzed (Participants) | 30
  Affective Problems T Score- Baseline | 59.2 (9.73)
  Affective Problems T Score- Month 12: number analyzed (Participants) | 21
  Affective Problems T Score- Month 12 | 57.5 (9.09)
  Affective Problems T Score- Month 24: number analyzed (Participants) | 6
  Affective Problems T Score- Month 24 | 59.3 (8.38)
  Affective Problems T Score- Study Exit: number analyzed (Participants) | 21
  Affective Problems T Score- Study Exit | 57.7 (9.13)
  Somatic Problems T Score- Baseline: number analyzed (Participants) | 28
  Somatic Problems T Score- Baseline | 55.6 (9.28)
  Somatic Problems T Score- Month 12: number analyzed (Participants) | 21
  Somatic Problems T Score- Month 12 | 54.3 (5.40)
  Somatic Problems T Score- Month 24: number analyzed (Participants) | 6
  Somatic Problems T Score- Month 24 | 54.8 (5.67)
  Somatic Problems T Score- Study Exit: number analyzed (Participants) | 20
  Somatic Problems T Score- Study Exit | 54.0 (5.25)
  Attention-Def. Hyp. Problems T Score- Baseline: number analyzed (Participants) | 29
  Attention-Def. Hyp. Problems T Score- Baseline | 60.3 (7.88)
  Attention-Def. Hyp. Problems T Score- Month 12: number analyzed (Participants) | 21
  Attention-Def. Hyp. Problems T Score- Month 12 | 60.5 (7.96)
  Attention-Def. Hyp. Problems T Score- Month 24: number analyzed (Participants) | 6
  Attention-Def. Hyp. Problems T Score- Month 24 | 67.2 (9.87)
  Attention-Def. Hyp. Problems T Score- Study Exit: number analyzed (Participants) | 21
  Attention-Def. Hyp. Problems T Score- Study Exit | 61.1 (8.60)
  Oppositional Defiant Problems T Score- Baseline: number analyzed (Participants) | 30
  Oppositional Defiant Problems T Score- Baseline | 57.1 (7.52)
  Oppositional Defiant Problems T Score- Month 12: number analyzed (Participants) | 21
  Oppositional Defiant Problems T Score- Month 12 | 55.8 (8.61)
  Oppositional Defiant Problems T Score- Month 24: number analyzed (Participants) | 6
  Oppositional Defiant Problems T Score- Month 24 | 56.3 (7.31)
  Oppositional Defiant Problems T Score- Study Exit: number analyzed (Participants) | 21
  Oppositional Defiant Problems T Score- Study Exit | 56.3 (8.60)
  Conduct Problems T Score- Baseline: number analyzed (Participants) | 28
  Conduct Problems T Score- Baseline | 56.4 (8.42)
  Conduct Problems T Score- Month 12: number analyzed (Participants) | 21
  Conduct Problems T Score- Month 12 | 54.7 (8.79)
  Conduct Problems T Score- Month 24: number analyzed (Participants) | 6
  Conduct Problems T Score- Month 24 | 55.7 (5.68)
  Conduct Problems T Score- Study Exit: number analyzed (Participants) | 20
  Conduct Problems T Score- Study Exit | 55.5 (8.23)
  Total Problems T Score- Baseline | 56.2 (12.00)
  Total Problems T Score- Month 12: number analyzed (Participants) | 21
  Total Problems T Score- Month 12 | 55.5 (10.20)
  Total Problems T Score- Month 24: number analyzed (Participants) | 6
  Total Problems T Score- Month 24 | 58.8 (6.85)
  Total Problems T Score- Study Exit: number analyzed (Participants) | 21
  Total Problems T Score- Study Exit | 56.1 (9.99)

7. Secondary Outcome: Mean Behavior Rating Inventory of Executive Function (BRIEF) Scores
Description: The Behavior Rating Inventory of Executive Function (BRIEF) is designed to assess executive functioning in children and adolescents ages 5 to 18 years of age. Parents/caregivers answered 86 questions on a 3-point scale (never, sometimes, often). Similar questions were grouped together into 8 scales; these scales were summed to produce 2 index measures and a global executive composite score. Raw scores for the indices/scales and composite score were converted to T-scores with corresponding 90% confidence intervals using computer software. Higher T-scores indicate a higher level of dysfunction.
Time Frame: Baseline, Month 12, Month 24, and study exit visit (up to 66 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | HPN-100- Pediatric
Number analyzed (Participants) | 30
T-Score
  Behavioral Regulation Index T Score- Baseline | 54.0 (9.58)
  Behavioral Regulation Index T Score- Month 12: number analyzed (Participants) | 21
  Behavioral Regulation Index T Score- Month 12 | 56.8 (10.96)
  Behavioral Regulation Index T Score- Month 24: number analyzed (Participants) | 7
  Behavioral Regulation Index T Score- Month 24 | 57.3 (8.54)
  Behavioral Regulation Index T Score- Study Exit: number analyzed (Participants) | 22
  Behavioral Regulation Index T Score- Study Exit | 56.1 (9.92)
  Metacognition Index T Score- Baseline | 57.7 (9.41)
  Metacognition Index T Score- Month 12: number analyzed (Participants) | 21
  Metacognition Index T Score- Month 12 | 59.0 (10.80)
  Metacognition Index T Score- Month 24: number analyzed (Participants) | 7
  Metacognition Index T Score- Month 24 | 61.3 (13.17)
  Metacognition Index T Score- Study Exit: number analyzed (Participants) | 22
  Metacognition Index T Score- Study Exit | 59.2 (10.20)
  Global Executive Composite T Score- Baseline | 56.7 (8.95)
  Global Executive Composite T Score- Month 12: number analyzed (Participants) | 21
  Global Executive Composite T Score- Month 12 | 58.7 (10.18)
  Global Executive Composite T Score- Month 24: number analyzed (Participants) | 7
  Global Executive Composite T Score- Month 24 | 60.6 (11.33)
  Global Executive Composite T Score- Study Exit: number analyzed (Participants) | 22
  Global Executive Composite T Score- Study Exit | 58.6 (9.52)

8. Secondary Outcome: Mean California Verbal Learning Test Scores: List A Total 1-5 T-Scores
Description: The California Verbal Learning Test - Second Edition (CVLT-II) assesses recall and recognition of word lists over several immediate- and delayed-memory trials. In the learning phase, adult participants were presented a list of 16 words (List A; 4 words each in 4 categories [e.g., fruit, toys, etc.]) for 5 trials, but words from the same category were never presented consecutively. An interference list (List B) of 16 different words was then presented for 1 trial. Short-and long-delay recalls for List A, yes/no recognition trials of List A, and a forced-choice recognition trial of List A was also administered. The total score for the 5 immediate-recall trials was converted to a T-score. Lower T-scores reflect worse performance.
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and study exit visit (up to 66 months)
Population: Adult participants (age 19-61) with available data; data were not analyzed for the 4 ongoing adult participants in Canada after the cutoff for the clinical study report (29 Oct 2015).
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | HPN-100 - Adult
Number analyzed (Participants) | 40
T-Score
  List A Total 1-5 T-Score- Baseline | 45.3 (13.80)
  List A Total 1-5 T-Score- Month 12: number analyzed (Participants) | 35
  List A Total 1-5 T-Score- Month 12 | 45.4 (14.83)
  List A Total 1-5 T-Score- Month 24: number analyzed (Participants) | 12
  List A Total 1-5 T-Score- Month 24 | 48.3 (17.67)
  List A Total 1-5 T-Score- Month 36: number analyzed (Participants) | 2
  List A Total 1-5 T-Score- Month 36 | 30.0 (22.63)
  List A Total 1-5 T-Score- Month 48: number analyzed (Participants) | 1
  List A Total 1-5 T-Score- Month 48 | 19.0
  List A Total 1-5 T-Score- Study Exit: number analyzed (Participants) | 36
  List A Total 1-5 T-Score- Study Exit | 46.3 (14.81)

9. Secondary Outcome: Mean California Verbal Learning Test Scores: Short and Long Delay Free Recall, Short and Long Delay Cued Recall, CVLT-II-Learning Slope, and Total Word Recognition Discrimination
Description: The California Verbal Learning Test - Second Edition (CVLT-II) assesses recall and recognition of word lists over several immediate- and delayed-memory trials. In the learning phase, adult participants were presented a list of 16 words (List A; 4 words each in 4 categories [e.g., fruit, toys, etc.]) for 5 trials, but words from the same category were never presented consecutively. An interference list (List B) of 16 different words was then presented for 1 trial. Short-and long-delay recalls for List A, yes/no recognition trials of List A, and a forced-choice recognition trial of List A was also administered. The scores for the learning slope, the short- and long-delay scores and total word recognition discrimination scores were converted to Z-scores by computer software. The CVLT-II Z-score has a mean of 0 and a standard deviation of 1. Negative scores indicate below-average performance.
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and study exit visit (up to 66 months)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | HPN-100 - Adult
Number analyzed (Participants) | 40
Z-Score
  Short Delay Free Recall Z Score- Baseline: number analyzed (Participants) | 39
  Short Delay Free Recall Z Score- Baseline | -0.6 (1.72)
  Short Delay Free Recall Z Score- Month 12: number analyzed (Participants) | 35
  Short Delay Free Recall Z Score- Month 12 | -0.4 (1.50)
  Short Delay Free Recall Z Score- Month 24: number analyzed (Participants) | 12
  Short Delay Free Recall Z Score- Month 24 | -0.6 (1.82)
  Short Delay Free Recall Z Score- Month 36: number analyzed (Participants) | 2
  Short Delay Free Recall Z Score- Month 36 | -2.0 (2.83)
  Short Delay Free Recall Z Score- Month 48: number analyzed (Participants) | 1
  Short Delay Free Recall Z Score- Month 48 | -3.5
  Short Delay Free Recall Z Score- Study Exit: number analyzed (Participants) | 36
  Short Delay Free Recall Z Score- Study Exit | -0.4 (1.47)
  Short Delay Cued Recall Z Score- Baseline: number analyzed (Participants) | 39
  Short Delay Cued Recall Z Score- Baseline | -0.6 (1.50)
  Short Delay Cued Recall Z Score- Month 12: number analyzed (Participants) | 35
  Short Delay Cued Recall Z Score- Month 12 | -0.4 (1.35)
  Short Delay Cued Recall Z Score- Month 24: number analyzed (Participants) | 12
  Short Delay Cued Recall Z Score- Month 24 | -0.2 (1.35)
  Short Delay Cued Recall Z Score- Month 36: number analyzed (Participants) | 2
  Short Delay Cued Recall Z Score- Month 36 | -1.8 (2.47)
  Short Delay Cued Recall Z Score- Month 48: number analyzed (Participants) | 1
  Short Delay Cued Recall Z Score- Month 48 | -4.0
  Short Delay Cued Recall Z Score- Study Exit: number analyzed (Participants) | 36
  Short Delay Cued Recall Z Score- Study Exit | -0.3 (1.37)
  Long Delay Free Recall Z Score- Baseline | -0.8 (1.72)
  Long Delay Free Recall Z Score- Month 12: number analyzed (Participants) | 35
  Long Delay Free Recall Z Score- Month 12 | -0.7 (1.61)
  Long Delay Free Recall Z Score- Month 24: number analyzed (Participants) | 12
  Long Delay Free Recall Z Score- Month 24 | -0.5 (2.12)
  Long Delay Free Recall Z Score- Month 36: number analyzed (Participants) | 2
  Long Delay Free Recall Z Score- Month 36 | -1.8 (3.18)
  Long Delay Free Recall Z Score- Month 48: number analyzed (Participants) | 1
  Long Delay Free Recall Z Score- Month 48 | -3.5
  Long Delay Free Recall Z Score- Study Exit: number analyzed (Participants) | 36
  Long Delay Free Recall Z Score- Study Exit | -0.5 (1.75)
  Long Delay Cued Recall Z Score- Baseline | -0.5 (1.50)
  Long Delay Cued Recall Z Score- Month 12: number analyzed (Participants) | 35
  Long Delay Cued Recall Z Score- Month 12 | -0.6 (1.62)
  Long Delay Cued Recall Z Score- Month 24: number analyzed (Participants) | 12
  Long Delay Cued Recall Z Score- Month 24 | -0.3 (1.75)
  Long Delay Cued Recall Z Score- Month 36: number analyzed (Participants) | 2
  Long Delay Cued Recall Z Score- Month 36 | -1.8 (2.47)
  Long Delay Cued Recall Z Score- Month 48: number analyzed (Participants) | 1
  Long Delay Cued Recall Z Score- Month 48 | -4.0
  Long Delay Cued Recall Z Score- Study Exit: number analyzed (Participants) | 36
  Long Delay Cued Recall Z Score- Study Exit | -0.4 (1.69)
  CVLT-II-Learning Slope Z Score- Baseline: number analyzed (Participants) | 39
  CVLT-II-Learning Slope Z Score- Baseline | -0.7 (1.15)
  CVLT-II-Learning Slope Z Score- Month 12: number analyzed (Participants) | 35
  CVLT-II-Learning Slope Z Score- Month 12 | -0.5 (1.51)
  CVLT-II-Learning Slope Z Score- Month 24: number analyzed (Participants) | 12
  CVLT-II-Learning Slope Z Score- Month 24 | -0.8 (1.34)
  CVLT-II-Learning Slope Z Score- Month 36: number analyzed (Participants) | 2
  CVLT-II-Learning Slope Z Score- Month 36 | -1.5 (1.41)
  CVLT-II-Learning Slope Z Score- Month 48: number analyzed (Participants) | 1
  CVLT-II-Learning Slope Z Score- Month 48 | -2.5
  CVLT-II-Learning Slope Z Score- Study Exit: number analyzed (Participants) | 36
  CVLT-II-Learning Slope Z Score- Study Exit | -0.8 (1.36)
  Total Recognition Discrim. Z Score- Baseline: number analyzed (Participants) | 39
  Total Recognition Discrim. Z Score- Baseline | -0.6 (1.48)
  Total Recognition Discrim. Z Score- Month 12: number analyzed (Participants) | 35
  Total Recognition Discrim. Z Score- Month 12 | -0.6 (1.39)
  Total Recognition Discrim. Z Score- Month 24: number analyzed (Participants) | 12
  Total Recognition Discrim. Z Score- Month 24 | -0.4 (2.00)
  Total Recognition Discrim. Z Score- Month 36: number analyzed (Participants) | 2
  Total Recognition Discrim. Z Score- Month 36 | -3.0 (2.12)
  Total Recognition Discrim. Z Score- Month 48: number analyzed (Participants) | 1
  Total Recognition Discrim. Z Score- Month 48 | -5.0
  Total Recognition Discrim. Z Score- Study Exit: number analyzed (Participants) | 36
  Total Recognition Discrim. Z Score- Study Exit | -0.6 (1.53)

ADVERSE EVENTS:
Time Frame: From the time of informed consent until 7 days after the last dose of study drug, up to 66 months
Arm/Group | HPN-100- Pediatric | HPN-100 - Adult
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 12/45 | 19/43
Other Adverse Events (participants affected / at risk) | 26/45 | 27/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100- Pediatric (N=45) | HPN-100 - Adult (N=43)
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Ammonia increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 10 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Psychological factor affecting medical condition (Psychiatric disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100- Pediatric (N=45) | HPN-100 - Adult (N=43)
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 6 | 5
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 3 | 2
Bronchitis (Infections and infestations) | 1 | 5
Ear infection (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 8
Amino acid level decreased (Investigations) | 3 | 0
Amino acid level increased (Investigations) | 3 | 1
Ammonia increased (Investigations) | 4 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Convulsion (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights.

DOCUMENTS (2):
  • Study Protocol (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT01257737/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT01257737/SAP_001.pdf